CLINICAL TRIAL: NCT01053663
Title: An Open-label, Prospective, Pharmacokinetic/Pharmacodynamic and Safety Evaluation of Intravenous Oseltamivir in the Treatment of Infants Less Than One Year of Age With Influenza Infection
Brief Title: A Study of Intravenous Oseltamivir [Tamiflu] in Infants With Influenza
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated prematurely after three influenza seasons.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP25138
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Results first posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-06

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Tamiflu

INTERVENTIONS:
Drug: Tamiflu — 10 doses over 5 or 6 days of which the first 5 or 6 doses must be intravenous, up to 5 days (10 doses) of additional intravenously or oral treatment if virus shedding continues at day 6

SUMMARY:
This open-label study will assess the pharmacokinetics and safety of oseltamivir [Tamiflu] in 3 cohorts of infants, aged 0-30 days, 31-90 days and 91-<365 days with influenza infection. Patients will receive 10 doses of intravenous oseltamivir [Tamiflu] therapy over 5 or 6 days. Optional oral therapy with oseltamivir [Tamiflu] may be considered following the intravenous dose associated with pharmacokinetic blood sampling. Evidence of continued virus shedding at day 6 can allow for up to 5 additional days (10 doses) of oral or intravenous administration. Anticipated time on study drug is 5-11 days. Target sample size is <50 patients.

ELIGIBILITY:
Inclusion Criteria:

* Infant patients
* Date of birth to date of enrollment is <1 year
* Diagnosis of influenza
* Duration of influenza symptoms </=96 hours prior to first dose
* - Parent/guardian willing to have patient receive intravenous therapy for 3 or 4 days (5 or 6 doses of study drug)

Exclusion Criteria:

* Date of conception to date of birth + date of birth to enrollment is <36 weeks
* Creatinine clearance <30 mL/min/1.73m2
* Patients receiving any form of renal replacement therapy at baseline
* Clinical evidence of severe hepatic decompensation at the time of enrollment
* Patients taking probenecid medication within 1 week prior to study day 1 or during the study

Max Age: 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (36):
- United States (35):
  - Little Rock, Arkansas
  - Los Angeles, California
  - Oakland, California
  - Orange, California
  - San Diego, California
  - Aurora, Colorado
  - Wilmington, Delaware
  - Jacksonville, Florida
  - Chicago, Illinois
  - South Bend, Indiana
  - Wichita, Kansas
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Omaha, Nebraska
  - Morristown, New Jersey
  - New Brunswick, New Jersey
  - Brooklyn, New York
  - New York, New York
  - Stony Brook, New York
  - Syracuse, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Toledo, Ohio
  - Providence, Rhode Island
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Richmond, Virginia
  - Madison, Wisconsin
- Petah Tikva, Israel

REFERENCES:
- [Derived] Munoz FM, Anderson EJ, Deville JG, Clinch B, Kamal MA. Pharmacokinetics and safety of intravenous oseltamivir in infants and children in open-label studies. Int J Clin Pharmacol Ther. 2015 Jul;53(7):531-40. doi: 10.5414/CP202307. PMID 26042486

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2428 participants were prescreened; of which, 2419 failed the prescreening evaluation. The most common reasons for failing the prescreening evaluation included the following: negative influenza diagnosis, not meeting the age criterion, ability to tolerate/absorb oral medication, and inability to comply with the study procedures.
Groups:
- Oseltamivir - All Participants: Participants received oseltamivir (Tamiflu) twice daily (every 12 hours) intravenously (IV) over 5 or 6 days for a total of 10 doses. The oseltamivir doses were based on participant's age. Participants aged 91 to less than (<) 365 days received 3 milligrams per kilogram (mg/kg); participants aged 31 to 90 days received 2.5 mg/kg; and participants aged 0 to 30 days received 2 mg/kg. For participants who did not receive all 10 doses IV, treatment could be completed with oral oseltamivir suspension (twice daily). If medically necessary, participants were allowed to receive an additional 10 doses of IV or oral oseltamivir after the initial 10 doses.
Period: Overall Study
Arm/Group | Oseltamivir - All Participants
Started | 9
Completed | 3
Not Completed | 6
Not completed — Death | 2
Not completed — Lost to Follow-up | 1
Not completed — Poor IV Access | 1
Not completed — Transferred to Another Hospital | 1
Not completed — Negative Influenza Diagnosis | 1

BASELINE CHARACTERISTICS:
Population: All-participants population included all participants who were enrolled in the study.
Groups:
- Oseltamivir: Age 91 to < 365 Days: Participants aged 91 to <365 days received oseltamivir 3 mg/kg twice daily (every 12 hours) IV over 5 or 6 days for a total of 10 doses. For participants who did not receive all 10 doses IV, treatment could be completed with oral oseltamivir suspension (twice daily). If medically necessary, participants were allowed to receive an additional 10 doses of IV or oral oseltamivir after the initial 10 doses.
- Oseltamivir: Age 31 to 90 Days: Participants aged 31 to 90 days received oseltamivir 2.5 mg/kg twice daily (every 12 hours) IV over 5 or 6 days for a total of 10 doses. For participants who did not receive all 10 doses IV, treatment could be completed with oral oseltamivir suspension (twice daily). If medically necessary, participants were allowed to receive an additional 10 doses of IV or oral oseltamivir after the initial 10 doses.
- Oseltamivir: Age 0 to 30 Days: Participants aged 0 to 30 days received oseltamivir 2 mg/kg twice daily (every 12 hours) IV over 5 or 6 days for a total of 10 doses. For participants who did not receive all 10 doses IV, treatment could be completed with oral oseltamivir suspension (twice daily). If medically necessary, participants were allowed to receive an additional 10 doses of IV or oral oseltamivir after the initial 10 doses.
- Total: Total of all reporting groups
Arm/Group | Oseltamivir: Age 91 to < 365 Days | Oseltamivir: Age 31 to 90 Days | Oseltamivir: Age 0 to 30 Days | Total
Number analyzed (Participants) | 7 | 1 | 1 | 9
Age, Continuous [Mean (Standard Deviation); unit: days] | 175.0 (62.0) | 41.0 | 23.0 | 143.2 (82.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 2
  Male | 5 | 1 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Versus Time Curve From Time Zero to Last Measurable Plasma Concentration (AUClast) of Oseltamivir and Oseltamivir Carboxylate on Day 1
Time Frame: Pre-dose (Hour 0), 2, 3-4, 5-7, and 10-12 hours post-dose on Day 1
Population: Pharmacokinetic (PK) population included all treated participants who had at least one blood sample evaluable for drug concentration level. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Oseltamivir: Age 91 to < 365 Days | Oseltamivir: Age 31 to 90 Days | Oseltamivir: Age 0 to 30 Days
Number analyzed (Participants) | 3 | 0 | 1
hour*nanogram/milliliter (h*ng/mL)
  Oseltamivir | 777 (162.8) |  | 494
  Oseltamivir Carboxylate | 5200 (87.8) |  | 7510

2. Primary Outcome: AUClast of Oseltamivir and Oseltamivir Carboxylate on Day 2
Time Frame: Pre-dose (Hour 0), 2, 3-4, 5-7, and 10-12 hours post-dose on Day 2
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Oseltamivir: Age 91 to < 365 Days | Oseltamivir: Age 31 to 90 Days | Oseltamivir: Age 0 to 30 Days
Number analyzed (Participants) | 3 | 1 | 0
h*ng/mL
  Oseltamivir | 988 (57.8) | 481 |
  Oseltamivir Carboxylate | 7270 (42.2) | 5330 |

3. Primary Outcome: AUClast of Oseltamivir and Oseltamivir Carboxylate on Day 4
Time Frame: Pre-dose (Hour 0), 2 and 4 hours post-dose on Day 4
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Oseltamivir: Age 91 to < 365 Days | Oseltamivir: Age 31 to 90 Days | Oseltamivir: Age 0 to 30 Days
Number analyzed (Participants) | 2 | 0 | 1
h*ng/mL
  Oseltamivir | 1520 (33.9) |  | 389
  Oseltamivir Carboxylate | 3880 (98.0) |  | 2070

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Oseltamivir and Oseltamivir Carboxylate on Day 1
Time Frame: Pre-dose (Hour 0), 2, 3-4, 5-7, and 10-12 hours post-dose on Day 1
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Oseltamivir: Age 91 to < 365 Days | Oseltamivir: Age 31 to 90 Days | Oseltamivir: Age 0 to 30 Days
Number analyzed (Participants) | 3 | 0 | 1
nanogram/milliliter (ng/mL)
  Oseltamivir | 307 (315.7) |  | 203
  Oseltamivir Carboxylate | 736 (55.5) |  | 871

5. Primary Outcome: Cmax of Oseltamivir and Oseltamivir Carboxylate on Day 2
Time Frame: Pre-dose (Hour 0), 2, 3-4, 5-7, and 10-12 hours post-dose on Day 2
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oseltamivir: Age 91 to < 365 Days | Oseltamivir: Age 31 to 90 Days | Oseltamivir: Age 0 to 30 Days
Number analyzed (Participants) | 3 | 1 | 0
ng/mL
  Oseltamivir | 419 (78.4) | 194 |
  Oseltamivir Carboxylate | 1080 (43.6) | 1050 |

6. Primary Outcome: Cmax of Oseltamivir and Oseltamivir Carboxylate on Day 4
Time Frame: Pre-dose (Hour 0), 2 and 4 hours post-dose on Day 4
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oseltamivir: Age 91 to < 365 Days | Oseltamivir: Age 31 to 90 Days | Oseltamivir: Age 0 to 30 Days
Number analyzed (Participants) | 2 | 0 | 1
ng/mL
  Oseltamivir | 742 (31.1) |  | 189
  Oseltamivir Carboxylate | 1370 (89.6) |  | 727

7. Secondary Outcome: Time to the Maximum Observed Plasma Concentration (Tmax) of Oseltamivir and Oseltamivir Carboxylate
Time Frame: Pre-dose (Hour 0), 2, 3-4, 5-7, and 10-12 hours post-dose on Day 1 and Day 2, pre-dose (Hour 0), 2 and 4 hours post-dose on Day 4
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome, n = number of participants evaluable for specified categories.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Oseltamivir: Age 91 to < 365 Days | Oseltamivir: Age 31 to 90 Days | Oseltamivir: Age 0 to 30 Days
Number analyzed (Participants) | 3 | 1 | 1
hours
  Day 1: Oseltamivir (n = 3, 0, 1) | 2.51 (55.4) | NA (NA) — Data not available as no participant was evaluable. | 2.00
  Day 1: Oseltamivir Carboxylate (n = 3, 0, 1) | 4.57 (32.5) | NA (NA) — Data not available as no participant was evaluable. | 5.58
  Day 2: Oseltamivir (n = 3, 1, 0) | 2.02 (1.4) | 2.13 | NA (NA) — Data not available as no participant was evaluable.
  Day 2: Oseltamivir Carboxylate (n = 3, 1, 0) | 3.40 (47.8) | 4.30 | NA (NA) — Data not available as no participant was evaluable.
  Day 4: Oseltamivir (n = 2, 0, 1) | 2.02 (1.2) | NA (NA) — Data not available as no participant was evaluable. | 1.93
  Day 4: Oseltamivir Carboxylate (n = 2, 0, 1) | 3.85 (6.7) | NA (NA) — Data not available as no participant was evaluable. | 3.98

8. Secondary Outcome: Last Measurable Plasma Concentration (Clast) of Oseltamivir and Oseltamivir Carboxylate
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oseltamivir: Age 91 to < 365 Days | Oseltamivir: Age 31 to 90 Days | Oseltamivir: Age 0 to 30 Days
Number analyzed (Participants) | 3 | 1 | 1
ng/mL
  Day 1: Oseltamivir (n = 3, 0, 1) | 5.58 (183.0) | NA (NA) — Data not available as no participant was evaluable. | 2.76
  Day 1: Oseltamivir Carboxylate (n = 3, 0, 1) | 505 (82.9) | NA (NA) — Data not available as no participant was evaluable. | 503
  Day 2: Oseltamivir (n = 3, 1, 0) | 8.22 (183.5) | 6.84 | NA (NA) — Data not available as no participant was evaluable.
  Day 2: Oseltamivir Carboxylate (n = 3, 1, 0) | 849 (67.9) | 948 | NA (NA) — Data not available as no participant was evaluable.
  Day 4: Oseltamivir (n = 2, 0, 1) | 66.2 (28.8) | NA (NA) — Data not available as no participant was evaluable. | 10.7
  Day 4: Oseltamivir Carboxylate (n = 2, 0, 1) | 1370 (89.6) | NA (NA) — Data not available as no participant was evaluable. | 727

9. Secondary Outcome: Time of the Last Measurable Plasma Concentration (Tlast) of Oseltamivir and Oseltamivir Carboxylate
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Oseltamivir: Age 91 to < 365 Days | Oseltamivir: Age 31 to 90 Days | Oseltamivir: Age 0 to 30 Days
Number analyzed (Participants) | 3 | 1 | 1
hours
  Day 1: Oseltamivir (n = 3, 0, 1) | 9.62 (24.7) | NA (NA) — Data not available as no participant was evaluable. | 10.58
  Day 1: Oseltamivir Carboxylate (n = 3, 0, 1) | 9.62 (24.7) | NA (NA) — Data not available as no participant was evaluable. | 10.58
  Day 2: Oseltamivir (n = 3, 1, 0) | 8.55 (51.1) | 6.47 | NA (NA) — Data not available as no participant was evaluable.
  Day 2: Oseltamivir Carboxylate (n = 3, 1, 0) | 8.55 (51.1) | 6.47 | NA (NA) — Data not available as no participant was evaluable.
  Day 4: Oseltamivir (n = 2, 0, 1) | 3.85 (6.7) | NA (NA) — Data not available as no participant was evaluable. | 3.98
  Day 4: Oseltamivir Carboxylate (n = 2, 0, 1) | 3.85 (6.7) | NA (NA) — Data not available as no participant was evaluable. | 3.98

10. Secondary Outcome: Number of Participants With Greater Than or Equal to (≥) 5-Fold Change in Neuraminidase Inhibition (NAI) Assay 50 Percent (%) Inhibitory Concentration (IC50) Values
Description: IC50 was defined as the concentration that causes 50% inhibition of viral activity. IC50 values were calculated using NAI assay. The 5-fold change was calculated as either ≥5 times change in the NAI IC50 visit value from the Reference value at a visit or ≥5 times change in the NAI IC50 Visit value from the Baseline value.
Time Frame: Baseline, Days 1, 3, 4, 6, 15
Population: Safety population included all participants who received at least one dose of IV study medication and had a safety assessment performed after initiation of treatment. Here, number of participants analyzed = participants evaluable for this outcome measure, and n = participants evaluable for specified time-point, for each arm, respectively.
Measure: Number; unit: participants
Groups:
- Oseltamivir: All Participants: Participants received oseltamivir twice daily (every 12 hours) IV over 5 or 6 days for a total of 10 doses. The oseltamivir doses were based on participant's age. Participants aged 91 to <365 days received 3 mg/kg; participants aged 31 to 90 days received 2.5 mg/kg; and participants aged 0 to 30 days received 2 mg/kg. For participants who did not receive all 10 doses IV, treatment could be completed with oral oseltamivir suspension (twice daily). If medically necessary, participants were allowed to receive an additional 10 doses of IV or oral oseltamivir after the initial 10 doses.
Arm/Group | Oseltamivir: Age 91 to < 365 Days | Oseltamivir: Age 31 to 90 Days | Oseltamivir: Age 0 to 30 Days | Oseltamivir: All Participants
Number analyzed (Participants) | 4 | 0 | 1 | 5
participants
  Day 1 (n=4, 0, 1, 5) | 1 |  | 0 | 1
  Day 3 (n=0, 0, 1, 1) | NA — Data not available as no participant was evaluable in this arm for specified time-point. |  | 0 | 0
  Day 4 (n=3, 0, 0, 3) | 1 |  | NA — Data not available as no participant was evaluable in this arm for specified time-point. | 1
  Day 6 (n=0, 0, 1, 1) | NA — Data not available as no participant was evaluable in this arm for specified time-point. |  | 0 | 0
  Day 15 (n=1, 0, 0, 1) | 0 |  | NA — Data not available as no participant was evaluable in this arm for specified time-point. | 0

11. Secondary Outcome: Number of Participants With Oseltamivir Resistance Mutation
Description: Resistance was assessed by neuraminidase (NA) and hemagglutinin (HA) genes sequencing analysis, using Reverse Transcription Polymerase Chain Reaction (RT-PCR).
Time Frame: Up to Day 30
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | Oseltamivir: Age 91 to < 365 Days | Oseltamivir: Age 31 to 90 Days | Oseltamivir: Age 0 to 30 Days | Oseltamivir: All Participants
Number analyzed (Participants) | 7 | 1 | 1 | 9
participants | 1 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to Day 30
Arm/Group | Oseltamivir: Age 91 to < 365 Days | Oseltamivir: Age 31 to 90 Days | Oseltamivir: Age 0 to 30 Days | Oseltamivir: All Participants
Serious Adverse Events (participants affected / at risk) | 5/7 | 0/1 | 0/1 | 5/9
Other Adverse Events (participants affected / at risk) | 4/7 | 0/1 | 1/1 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oseltamivir: Age 91 to < 365 Days (N=7) | Oseltamivir: Age 31 to 90 Days (N=1) | Oseltamivir: Age 0 to 30 Days (N=1) | Oseltamivir: All Participants (N=9)
Multi-Organ Failure (General disorders) | 1 | 0 | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 1 | 0 | 0 | 1
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oseltamivir: Age 91 to < 365 Days (N=7) | Oseltamivir: Age 31 to 90 Days (N=1) | Oseltamivir: Age 0 to 30 Days (N=1) | Oseltamivir: All Participants (N=9)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Application Site Vesicles (General disorders) | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Brain Oedema (Nervous system disorders) | 1 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Low number of participants enrolled in the study at the time that the study was terminated limits conclusions that can be derived from the study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.